CLINICAL TRIAL: NCT02496416
Title: Comparison of Two Physical Activity Interventions in Individuals With Multiple Sclerosis: A Randomized Clinical Trial
Brief Title: Comparison of Two Physical Activity Interventions in Individuals With Multiple Sclerosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kessler Foundation (Other)
Collaborators: National Multiple Sclerosis Society (Other)
Responsible Party: Principal Investigator, Helen Genova, Research Scientist, Kessler Foundation
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: R-876-15
Record Dates: First submitted 2015-07-07; First posted 2015-07-14 (Estimated); Last update posted 2022-12-05 (Actual); Status verified 2022-12

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment (Experimental): The treatment group will participate in an eight week aquatic exercise program during weeks 2-9 of the study. The aquatic exercise program will consist of 45 minute classes held 3 days/week for 8 weeks (18 hours total). The program is based on guidelines provided by the National Multiple Sclerosis Society (NMSS) and will be led by an aquatic fitness instructor certified to teach individuals with MS at the YMCA in Randolph, NJ.. The exercises will focus on improving flexibility, balance and strength. Equipment such as water mitts, paddles, noodles and bands will be used to increase the level of difficulty as needed.
  Interventions: Behavioral: Aquatic Exercise Program
- Control (Active Comparator): The control group will participate in an eight week stretching program during weeks 2-9 of the study. The stretching program will consist of 45 minute classes held 3 days/week for 8 weeks (18 hours total). The program is based on guidelines provided by the National Multiple Sclerosis Society (NMSS) and will be conducted online via a secure video-conferencing website.
  Interventions: Behavioral: Stretching Program

INTERVENTIONS:
Behavioral: Aquatic Exercise Program — The aquatic exercise program will consist of 45 minute classes held 3 days/week for 8 weeks (18 hours total). The program is based on guidelines provided by the National Multiple Sclerosis Society (NMSS) and will be led by an aquatic fitness instructor certified to teach individuals with MS at the YMCA in Scotch Plains-Fanwood. The exercises will focus on improving flexibility, balance and strength. Equipment such as water mitts, paddles, noodles and bands will be used to increase the level of difficulty as needed.
  Arms: Treatment
Behavioral: Stretching Program — The stretching program will consist of 45 minute classes held 3 days/week for 8 weeks (18 hours total). The program is based on guidelines provided by the National Multiple Sclerosis Society (NMSS) and will be conducted online via a secure video-conferencing website.
  Arms: Control

SUMMARY:
This study will examine the effectiveness of aquatic therapy on a range of MS-related symptoms such as cognition, mood, fatigue and quality of life (QOL).

DETAILED DESCRIPTION:
Aim 1. Examine the impact of aquatic exercise on cognitive abilities. The proposed study will test the hypotheses that, compared to the wait-list control group, the treatment group will demonstrate significantly greater improvements in cognitive outcomes, specifically: processing speed, executive functioning, working memory and long-term memory.

Aim 2. The current study will examine the impact of an aquatic exercise on fatigue, mood, wellness, QOL and physical functioning. Specifically the investigators predict that aquatic exercise will lead to improvements in: 1.Fatigue 2. Health related QOL 3. Depression/anxiety 4. Self-efficacy 5. Physical Functioning (i.e. gait and walking).

Aim 3: Examine the long-term effects of aquatic exercise on all outcome measures.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of MS.
* between the ages of 18-65.
* read and speak English fluently.

Exclusion Criteria:

* history of significant substance abuse.
* history of neurological disease other than MS (for example, stroke, epilepsy, or brain injury).
* history of significant psychiatric illness (for example, bipolar disorder or schizophrenia).
* has engaged in more than 30 minutes of moderate to strenuous exercise per week during the past six months.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-08 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Cognition measured by results of standardized neuropsychological tests | 8 weeks
  standardized measures of processing speed, executive functioning, working memory and long-term memory

SECONDARY OUTCOMES:
Fatigue measured by self-report questionnaires | 8 weeks
  Modified Fatigue Impact Scale (MFIS) and Fatigue Severity Scale (FSS_
Quality of Life measured by self report questionnaires | 8 weeks
  General QOL measured with Satisfaction with Life Scale (SWLS) and HRQOL measured with Health Status Questionnaire (HSQ).

CONTACTS AND LOCATIONS:
Overall Officials: Helen Genova, PhD, Principal Investigator — Kessler Foundation
Locations (1):
- Kessler Foundation, East Hanover, New Jersey, United States